CLINICAL TRIAL: NCT00866840
Title: A Phase II Trial of Riluzole in Patients With Advanced Melanoma
Brief Title: Riluzole in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0220080280; P30CA072720 (NIH); CINJ-090802 (Other: CINJ); CDR0000637646 (Other: CDR)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Riluzole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riluzole (Experimental): 100 mg orally twice daily
  Interventions: Drug: riluzole

INTERVENTIONS:
Drug: riluzole — 100 mg orally twice daily

SUMMARY:
RATIONALE: Riluzole may stop or slow the growth of tumor cells and may be an effective treatment for melanoma.

PURPOSE: This phase II trial is studying how well riluzole works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether administration of a daily dose of riluzole results in tumor shrinkage, as measured by RECIST criteria, in patients with advanced melanoma.

Secondary

* Determine the long-term toxicity of riluzole when administered to these patients.
* Compare the survival of these patients with historical controls.

OUTLINE: Patients receive oral riluzole twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Unresectable stage III or stage IV disease
* Measurable disease according to RECIST criteria, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques or > 10 mm by spiral CT scan
* No known brain metastases unless treated and stable for ≥ 2 weeks by MRI evaluation

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 50,000/μL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST/ALT ≤ 3 times ULN
* INR ≤ 1.5 times ULN
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 weeks after completion of study treatment
* No second primary malignancy, except carcinoma in situ of the cervix, adequately treated nonmelanoma carcinoma of the skin, or other malignancy treated ≥ 5 years ago with no evidence of recurrence
* No concurrent serious systemic disorders (including active infections) that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* No history of allergic reactions attributed to riluzole
* No known history of hepatitis B or C

PRIOR CONCURRENT THERAPY:

* No more than 1 prior therapeutic chemotherapy regimen for advanced melanoma
* Prior treatment with riluzole on clinical trial CINJ-090603 allowed
* No other concurrent investigational or commercial agents or therapies for the treatment of the malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James S. Goydos, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mehnert JM, Silk AW, Lee JH, Dudek L, Jeong BS, Li J, Schenkel JM, Sadimin E, Kane M, Lin H, Shih WJ, Zloza A, Chen S, Goydos JS. A phase II trial of riluzole, an antagonist of metabotropic glutamate receptor 1 (GRM1) signaling, in patients with advanced melanoma. Pigment Cell Melanoma Res. 2018 Jul;31(4):534-540. doi: 10.1111/pcmr.12694. Epub 2018 Apr 10. PMID 29453787

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riluzole
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Riluzole
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response as Measured by RECIST Criteria
Description: Per Response Evaluation Criteria in Solid Tumors (RECIST v1.0) for target lesions and assessed by CT or MRI imaging: Complete response (CR) - disappearance of all target lesions; Partial response (PR) - >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) - At least a 20% increase in the sum of the longest diameter of target lesions; or Stable Disease (SD) - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Imaging for tumor assessments was performed after 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole
Number analyzed (Participants) | 13
Participants
  Stable disease | 6
  Progressive disease | 7
Statistical Analysis 1: Comparison: Riluzole; No objective responses were seen in the first phase and accrual was stopped; Test type: Other; No objective responses were seen in the first phase and accrual was stopped

2. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: Adverse events (AEs) were evaluated and graded using the National Cancer Institute Common Toxicity Criteria, version 3.0.
Time Frame: From date of randomization through completion of follow-up, up to three years
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole
Number analyzed (Participants) | 13
Participants | 9

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier plots of probability of overall survival.
Time Frame: Overall survival at one year
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole
Number analyzed (Participants) | 13
Participants | 1

ADVERSE EVENTS:
Time Frame: From date of randomization through completion of follow-up, up to three years
Arm/Group | Riluzole
All-Cause Mortality (participants affected / at risk) | 4/13
Serious Adverse Events (participants affected / at risk) | 10/13
Other Adverse Events (participants affected / at risk) | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=13)
Dizziness (General disorders) | 1 (2)
Muscle weakness, generalized or specific area (General disorders) | 2 (2) — (not due to neuropathy) - Extremity-upper
Death (General disorders) | 1 (1) — not associated with CTCAE term - Disease progression NOS
Infection (Infections and infestations) | 1 (1) — with normal ANC or Grade 1 or 2 neutrophils - Abdomen NOS
Dehydration (General disorders) | 2 (2)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 1 (1) — left arm
Neuropathy: motor (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=13)
Gastrointestinal (Gastrointestinal disorders) | 7 (11)
Constitutional Symptoms (Gastrointestinal disorders) | 8 (10)
Neurology (Nervous system disorders) | 7 (14)
Pain (General disorders) | 5 (7)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 3 (10)
Musculoskeletal/Soft Tissue (Musculoskeletal and connective tissue disorders) | 3 (3)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 2 (2)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cardiac General (Cardiac disorders) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Ocular/Visual (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes